CLINICAL TRIAL: NCT02164448
Title: The Effects of Intraoperative Dexmedetomidine Infusion on Postoperative Bowel Movement in Patients Undergoing Laparoscopic Gastrectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 4-2014-0249
Record Dates: First submitted 2014-06-09; First posted 2014-06-16 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Gastric Cancer Patients Undergoing Laparoscopic Gastrectomy
Keywords: dexmedetomidine; postoperative bowel movement; laparoscopic gastrectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexmedetomidine group (Experimental)
  Interventions: Drug: the dexmedetomidine group
- control group (Placebo Comparator)
  Interventions: Drug: the control group

INTERVENTIONS:
Drug: the dexmedetomidine group — the dexmedetomidine group: dexmedetomidine infusion from induction of anesthesia to end of surgery
  Arms: dexmedetomidine group
Drug: the control group — saline infusion from induction of anesthesia to end of surgery
  Arms: control group

SUMMARY:
The investigators hypothesized that sympatholytic effect of dexmedetomidine would attenuate the hemodynamic instability and decrease in the splanchnic blood flow caused by pneumoperitoneum during laparoscopic surgery. This study is to investigate the effect of intraoperative dexmedetomidine infusion on postoperative bowel movement in patients undergoing laparoscopic gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

* patient between 20 and 65 of age with ASA physical status Ⅰ-Ⅲ
* gastric cancer patient undergoing laparoscopic gastrectomy

Exclusion Criteria:

* ASA physical status Ⅳ
* bradycardia (< 60 bpm), arrhythmia
* uncompensated heart failure
* hepatic failure (Child-Pugh score B 이상)
* renal failure (eGFR MDRD < 60 ml/min/1.73m2)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
gas passing | up to 1 week
  To evaluate the postoperative bowel movement, we will assess the time to first gas passing

SECONDARY OUTCOMES:
sips of water time | up to 1 week
  To evaluate the postoperative bowel movement, we will assess the time to resume water intake

OTHER OUTCOMES:
soft diet time | up to 1 week
  To evaluate the postoperative bowel movement, we will assess the time to resume soft diet intake

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine,, Seoul, Seoul, South Korea